CLINICAL TRIAL: NCT04496921
Title: Vitamin K Supplementation to Reduce Deficiencies in Adults With Cystic Fibrosis : A Pilot Study
Brief Title: Vitamin K Supplementation to Reduce Deficiencies in Adults With Cystic Fibrosis
Acronym: VITK-FK
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical care of patients with CF changed following COVID-19 pandemic (OGTT not performed at the CF clinic since March 2020); in consequence, this study is no longer feasible.
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VITK-FK
Record Dates: First submitted 2020-07-21; First posted 2020-08-04 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis
Keywords: Vitamin K; Supplementation; Nutrition; Diabetes
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: * Group A: vitamin K supplement of 2 mg, once a day for 6 months
  * Group B: vitamin K supplement of 7 mg, twice a week for 6 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin K supplement, dose #1 (Active Comparator): Vitamin K supplementation with dose #1
  Interventions: Dietary Supplement: Vitamin K supplementation, dose #1
- Vitamin K supplement, dose #2 (Active Comparator): Vitamin K supplementation with dose #2
  Interventions: Dietary Supplement: Vitamin K supplementation, dose #2

INTERVENTIONS:
Dietary Supplement: Vitamin K supplementation, dose #1 — Vitamin K supplement : 2mg, once a day, for 6 months. Complete biochemical profile, weight and size (body mass index), drugs list, pulmonary function by spirometry (FEV, etc.). Food frequency questionnaire.
  Arms: Vitamin K supplement, dose #1
Dietary Supplement: Vitamin K supplementation, dose #2 — Vitamin K supplement : 7mg, twice a week, for 6 months. Complete biochemical profile, weight and size (body mass index), drugs list, pulmonary function by spirometry (FEV, etc.). Food frequency questionnaire.
  Arms: Vitamin K supplement, dose #2

SUMMARY:
Cystic fibrosis (CF) patients are at risk for vitamin K deficiencies. Supplementation for fat-soluble vitamins A, D, and E is well established, but in CF, there is little data for vitamin K concerning the optimal dose and frequency of supplementation. Beyond its known role in coagulation, research has highlighted the role of vitamin K for bone health and the control of blood sugar levels. However, after pulmonary complications, the risk of diabetes and bone diseases are two important and frequent complications of CF. Patients with CF being at risk of vitamin K deficiencies, this vitamin could play a role in these complications.

DETAILED DESCRIPTION:
The investigators propose a pilot study (carried out to assess its feasibility on a larger scale) to evaluate if a supplement of vitamin K improves vitamin K serum levels in CF patients by comparing:

* Group A: a vitamin K supplement of 2mg, every day for 6 months
* Group B: a vitamin K supplement of 7mg, twice a week for 6 months

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CF
* Aged above 18 years
* Pancreatic insufficient
* Subjects with an OGTT test in the last 12 months or subjects who are diabetic

Exclusion Criteria:

* Receive or have received, in the last 6 months, a supplement of vitamin K (dose greater than 500 mcg per day)
* Subjects with a pulmonary function under 30%
* Subjects with severe gastrointestinal disease (Crohn disease, coeliac disease and recent (<1 year) history of intestinal occlusion).
* Subjects with a history of liver disease (severe or transplant)
* Known allergy or intolerance to phylloquinone (oral form of vitamin K)
* Pregnancy (current or planned in the next 6 months)
* Subjects with signs of active secondary infections should wait at least 1 month after the end of antibiotic treatment in order to be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Change in serum vitamin K levels from baseline at 6 months | 0, 3 and 6 months
  Impact of supplementation on vitamin K serum levels

SECONDARY OUTCOMES:
Change in osteocalcin levels from baseline at 6 months | 0, 3 and 6 months
  Impact of supplementation on osteocalcin levels (Total and uncarboxylated)
Patient's perception and side effects of the supplement | 6 months
  Visual analogue scale questionnaire
Bone marker levels | 0, 3 and 6 months
  Impact of supplementation on bone marker C-Telopeptide
Glycemic marker levels | 0, 3 and 6 months
  Impact of supplementation on HbA1c levels and fructosamine levels

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Montreal Clinical Research Institute
Locations (2):
- Canada (2):
  - Montreal Clinical Research Institute (IRCM), Montreal, Quebec
  - CHUM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No